CLINICAL TRIAL: NCT05296044
Title: This Study Evaluates the Addition of Dapagliflozin in the Treatment of Type 2 Diates With Metformin and JT-003 Combination Therapy.
Brief Title: To Evaluate the Efficacy and Safety of JT-003 add-on in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin and Dapagliflozin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JLP-2008-302
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JT-003 (Experimental): Drug: JT-003
  Interventions: Drug: JT-003
- JT-003 Placebo (Placebo Comparator): Drug: JT-003 Placebo
  Interventions: Drug: JT-003 Placebo

INTERVENTIONS:
Drug: JT-003 — Subjects take the investigational products once a day for 24 weeks.
  Arms: JT-003
Drug: JT-003 Placebo — Subjects take the investigational products once a day for 24 weeks.
  Arms: JT-003 Placebo

SUMMARY:
A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of JT-003 Add-on in Patients with Type 2 Diabetes Mellitus Inadequately Controlled with Metformin and Dapagliflozin

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older with type 2 diabetes mellitus
2. Subjects with 7.0% ≤ HbA1c ≤ 11% at baseline
3. Those with > 45 kg/m2 of BMI
4. Those who voluntarily signed the informed consent to participate in this study

Exclusion Criteria:

1. Those who had allergic reaction to main ingredients or components of the investigational products.
2. Patients with the following major systemic disease

   * Patients with type 1 diabetes mellitus, secondary diabetes, or congenital renal diabetes etc.)
   * Patients with pituitary insufficiency or adrenal dysfunction
   * Patients with uncontrolled glycosemia(FPG > 270 mg/dL)
   * Patients with uncontrolled hypertension(SBP > 180 mmHg or DBP > 110 mmHg
   * Patients with severe hypertriglyceridemia (Triglyceride > 500 mg/dL)
   * Patients with severe renal dysfunction
   * Patients with liver dysfunction
   * Patients with AIDS
   * Those with clinically significant severe infection or trauma based on an investigator's judgement
   * Patients with pulmonary infarction, severe pulmonary dysfunction, hypoxemia
   * Unstable mental illness not regulated by drugs
   * Those who suffered from gastrointestinal diseases that may affect the absorption, distribution, metabolism, and excretion of investigational products or had underwent surgery;
   * Those who had genetic disorders such as galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption
3. Those with a history of malignant tumor within 5 years
4. Those with history of alcohol or drug abuse within 1 years
5. Those with heart failure (NYHA class II~IV) or who had suffered from heart failure within 6 months
6. Those who underwent surgery requiring general anesthesia within 4 weeks as of Visit 1 or who are scheduled to receive such surgery within 4 weeks after the study ends
7. Those who need to take prohibited concomitant medications stated during the study period.
8. Females who are pregnant or breastfeeding or patients planning to become pregnant or of childbearing potential, but not using any recognized contraceptive method
9. Those who are judged unsuitable for the study by a principal investigator or investigators
10. Those who have been administered with the following drugs or expected to require the continued administration during the study period:

    * Those who have been administered with obesity drugs within 12 weeks
    * Those being administered with thyroid medications and whose dose has been modified within 6 weeks
    * Those administered with systemic steroid agents (Prednisolone, >30 mg/day) within 2 weeks
    * Those being administered with diuretics and whose dose has been modified within 8 weeks as (however, dose reduction is accepted.)
11. Those who are currently participating in other ongoing clinical studies or those who have taken the investigational products from other clinical studies within 12 weeks

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2022-04-05 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1c | 24 week from the baseline
  Changes in HbA1c at the 24 week from the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Hong JH, Han KA, Hwang YC, Hong EG, Kim HJ, Lee CB, Cho HC, Won JC, Kim HS, Kim EH, Koh G, Ahn KH, Park KS. Efficacy and Safety of High-Dose Pioglitazone as Add-on Therapy in Patients with Type 2 Diabetes Mellitus Inadequately Controlled with Dapagliflozin and Metformin: Double-Blind, Randomized, Placebo-Controlled Trial. Diabetes Metab J. 2025 Oct 28. doi: 10.4093/dmj.2024.0696. Online ahead of print. PMID 41151541